CLINICAL TRIAL: NCT03242018
Title: A Randomized, Double-blind, Placebo-controlled, 3-arm, Parallel-group 52-week Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin in Patients With Type 2 Diabetes Mellitus and Severe Renal Impairment Who Have Inadequate Glycemic Control
Brief Title: A Study to Evaluate Safety and Effects of Sotagliflozin 400 and 200 mg on Glucose Control in Participants With Type 2 Diabetes, Severe Impairment of Kidney Function and Inadequate Blood Sugar Control
Acronym: SOTA-CKD4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15166; 2016-004906-32; U1111-1190-7589 (Other: UTN)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease Stage 4
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Following a 2-week run-in phase, participants received two placebo tablets (identical to sotagliflozin 200 milligrams [mg] in appearance) orally once daily for up to 56 weeks.
  Interventions: Drug: Placebo
- Sotagliflozin 200 mg (Experimental): Following a 2-week run-in phase, participants received two tablets, one sotagliflozin 200 mg tablet and one placebo tablet (identical to sotagliflozin 200 mg in appearance), orally once daily for up to 56 weeks.
  Interventions: Drug: Placebo; Drug: Sotagliflozin
- Sotagliflozin 400 mg (Experimental): Following a 2-week run-in phase, participants received sotagliflozin 400 mg, administered as 2 sotagliflozin 200 mg tablets, orally once daily for up to 56 weeks.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Placebo — Placebo tablet (identical to sotagliflozin 200 mg in appearance) orally, once daily.
  Arms: Placebo; Sotagliflozin 200 mg
Drug: Sotagliflozin — Sotagliflozin 200 mg, tablet, orally, once daily.
  Other Names: SAR439954
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg

SUMMARY:
Primary Objective:

To demonstrate the superiority of sotagliflozin 400 milligrams (mg) versus placebo with respect to hemoglobin A1c (HbA1c) reduction at Week 26 in participants with Type 2 diabetes who have inadequate glycemic control and severe renal impairment

Secondary Objectives:

* To assess the effects of sotagliflozin 200 mg versus placebo based on change from baseline in HbA1c
* To assess the effects of sotagloflozin 400 mg and 200 mg versus placebo
* To evaluate the safety of sotagliflozin 400 mg and 200 mg versus placebo

DETAILED DESCRIPTION:
The study duration is up to 60 weeks including 4 weeks prior to randomization, 52 weeks of randomized treatment and a visit 4 weeks after completion of the randomized treatment period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes (drug-naïve or on antidiabetic therapy) and documented severe renal insufficiency - CKD4 - defined by an estimated glomerular filtration rate (eGFR) equation (based on the 4 variable modification of diet in renal disease (MDRD) equation) of ≥15 and <30 milliliter per minute (mL/min)/1.73 per meter square (m^2).
* Signed written informed consent to participate in the study in accordance with local regulations.

Exclusion criteria:

* At the time of screening, age <18 years.
* Hemoglobin A1c (HbA1c) <7% or >11%.
* Type 1 diabetes.
* Women of childbearing potential (WOCBP) not willing to use highly effective method(s) of birth control during the study treatment period and the follow-up period, or who are unwilling or unable to be tested for pregnancy during the study.
* Treatment with an sodium-glucose cotransporter type 2 (SGLT2) inhibitor (canagliflozin, dapagliflozin, empagliflozin) during the last 12 months.
* Uncontrolled high blood pressure, severe anemia, severe cardiovascular problems, such as heart failure, active cancer, or other conditions that the Investigator believes with result in a short life expectancy, will preclude their safe participation in this study, or will make implementation of the protocol or interpretation of the study results difficult.
* Lower extremity complications (such as skin ulcers, infection, osteomyelitis and gangrene) identified during the Screening period, and still requiring treatment at Randomization.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (106):
- United States (34):
  - Investigational Site Number 8405033, Guntersville, Alabama
  - Investigational Site Number 8405005, Phoenix, Arizona
  - Investigational Site Number 8405007, Little Rock, Arkansas
  - Investigational Site Number 8405015, Chula Vista, California
  - Investigational Site Number 8405032, La Jolla, California
  - Investigational Site Number 8405003, Norco, California
  - Investigational Site Number 8405013, Northridge, California
  - Investigational Site Number 8405018, San Dimas, California
  - Investigational Site Number 8405021, Clearwater, Florida
  - Investigational Site Number 8405001, DeLand, Florida
  - Investigational Site Number 8405043, Miami, Florida
  - Investigational Site Number 8405006, Ocoee, Florida
  - Investigational Site Number 8405025, Ormond Beach, Florida
  - Investigational Site Number 8405039, Lawrenceville, Georgia
  - Investigational Site Number 8405041, Arlington Heights, Illinois
  - Investigational Site Number 8405030, Sellersburg, Indiana
  - Investigational Site Number 8405019, Lake Charles, Louisiana
  - Investigational Site Number 8405034, Flint, Michigan
  - Investigational Site Number 8405012, Norfolk, Nebraska
  - Investigational Site Number 8405035, Albany, New York
  - Investigational Site Number 8405027, Laurelton, New York
  - Investigational Site Number 8405014, The Bronx, New York
  - Investigational Site Number 8405037, New Bern, North Carolina
  - Investigational Site Number 8405038, Winston-Salem, North Carolina
  - Investigational Site Number 8405009, Dayton, Ohio
  - Investigational Site Number 8405004, Beaumont, Texas
  - Investigational Site Number 8405036, Dallas, Texas
  - Investigational Site Number 8405020, Houston, Texas
  - Investigational Site Number 8405026, Houston, Texas
  - Investigational Site Number 8405047, Hurst, Texas
  - Investigational Site Number 8405031, San Antonio, Texas
  - Investigational Site Number 8405016, San Antonio, Texas
  - Investigational Site Number 8405008, Layton, Utah
  - Investigational Site Number 8405040, Winchester, Virginia
- Argentina (3):
  - Investigational Site Number 0325001, Buenos Aires
  - Investigational Site Number 0325003, Launs Este
  - Investigational Site Number 0325004, Mar del Plata
- Brazil (4):
  - Investigational Site Number 0765003, Belém
  - Investigational Site Number 0765001, Fortaleza
  - Investigational Site Number 0765004, Rio de Janeiro
  - Investigational Site Number 0765002, São Paulo
- Colombia (4):
  - Investigational Site Number 1705004, Barranquilla
  - Investigational Site Number 1705005, Bogotá
  - Investigational Site Number 1705002, Manizales
  - Investigational Site Number 1705001, Zipaquirá
- Germany (3):
  - Investigational Site Number 2765001, Frankfurt am Main
  - Investigational Site Number 2765003, Hanover
  - Investigational Site Number 2765004, Münster
- Hungary (3):
  - Investigational Site Number 3485005, Baja
  - Investigational Site Number 3485007, Debrecen
  - Investigational Site Number 3485004, Pécs
- Israel (7):
  - Investigational Site Number 3765002, Ashkelon
  - Investigational Site Number 3765001, Haifa
  - Investigational Site Number 3765007, Kfar Saba
  - Investigational Site Number 3765005, Ramat Gan
  - Investigational Site Number 3765004, Rehovot
  - Investigational Site Number 3765006, Safed
  - Investigational Site Number 3765003, Tel Aviv
- Italy (6):
  - Investigational Site Number 3805003, Catania
  - Investigational Site Number 3805005, Milan
  - Investigational Site Number 3805006, Napoli
  - Investigational Site Number 3805002, Napoli
  - Investigational Site Number 3805001, Pavia
  - Investigational Site Number 3805004, Roma
- Mexico (8):
  - Investigational Site Number 4845001, Guadalajara
  - Investigational Site Number 4845004, Guadalajara
  - Investigational Site Number 4845007, Guadalajara Jalisco
  - Investigational Site Number 4845008, Merida, Yucatan
  - Investigational Site Number 4845006, Monterrey, N.L
  - Investigational Site Number 4845003, Morelia
  - Investigational Site Number 4845002, Querétaro
  - Investigational Site Number 4845005, Xalapa
- Poland (5):
  - Investigational Site Number 6165003, Krakow
  - Investigational Site Number 6165002, Lodz
  - Investigational Site Number 6165004, Oświęcim
  - Investigational Site Number 6165005, Puławy
  - Investigational Site Number 6165001, Rzeszów
- Romania (6):
  - Investigational Site Number 6425005, Bacau
  - Investigational Site Number 6425002, Bucharest
  - Investigational Site Number 6425003, Bucharest
  - Investigational Site Number 6425007, Hunedoara
  - Investigational Site Number 6425004, Lasi
  - Investigational Site Number 6425001, Târgu Mureş
- Russia (5):
  - Investigational Site Number 6435004, Chelyabinsk
  - Investigational Site Number 6435005, Kemerovo
  - Investigational Site Number 6435003, Krasnodar
  - Investigational Site Number 6435006, Novosibirsk
  - Investigational Site Number 6435001, Saint Petersburg
- South Africa (4):
  - Investigational Site Number 7105003, Cape Town
  - Investigational Site Number 7105004, Cape Town
  - Investigational Site Number 7105001, Johannesburg
  - Investigational Site Number 7105002, Pretoria
- Spain (8):
  - Investigational Site Number 7245005, Barcelona
  - Investigational Site Number 7245007, Barcelona
  - Investigational Site Number 7245003, Ferrol
  - Investigational Site Number 7245009, Granada
  - Investigational Site Number 7245006, Madrid
  - Investigational Site Number 7245004, Málaga
  - Investigational Site Number 7245001, Seville
  - Investigational Site Number 7245002, Zaragoza
- Ukraine (6):
  - Investigational Site Number 8045004, Chernivtsi
  - Investigational Site Number 8045006, Kiev
  - Investigational Site Number 8045007, Kyiv
  - Investigational Site Number 8045003, Kyiv
  - Investigational Site Number 8045001, Kyiv
  - Investigational Site Number 8045002, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Cherney DZI, Ferrannini E, Umpierrez GE, Peters AL, Rosenstock J, Carroll AK, Lapuerta P, Banks P, Agarwal R. Efficacy and safety of sotagliflozin in patients with type 2 diabetes and severe renal impairment. Diabetes Obes Metab. 2021 Dec;23(12):2632-2642. doi: 10.1111/dom.14513. Epub 2021 Aug 20. PMID 34338408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 106 investigative sites in United States, Argentina, Brazil, Colombia, Germany, Hungary, Israel, Italy, Mexico, Poland, Romania, Russian Federation, South Africa, Spain, Ukraine from 16 August 2017 to 11 December 2019.
Pre-assignment Details: A total of 277 participants with a diagnosis of Type 2 Diabetes Mellitus were randomized 1:1:1 to 1 of the 3 treatment groups: Placebo, Sotagliflozin 200 milligram (mg) and Sotagliflozin 400 mg.
Groups:
- Placebo: Following a 2-week run-in phase, participants received two placebo tablets (identical to sotagliflozin 200 mg in appearance) orally once daily for up to 56.3 weeks.
- Sotagliflozin 200 mg: Following a 2-week run-in phase, participants received two tablets, one sotagliflozin 200 mg tablet and one placebo tablet (identical to sotagliflozin 200 mg in appearance), orally once daily for up to 55.3 weeks.
- Sotagliflozin 400 mg: Following a 2-week run-in phase, participants received sotagliflozin 400 mg, administered as 2 sotagliflozin 200 mg tablets, orally once daily for up to 56.1 weeks.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 93 | 92 | 92
Completed | 75 | 78 | 78
Not Completed | 18 | 14 | 14
Not completed — Adverse Event | 7 | 7 | 6
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — At the Participant's Own Request | 5 | 1 | 4
Not completed — Reason Not Specified | 3 | 4 | 1
Not completed — Study Terminated by Sponsor | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 93 | 92 | 92 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.3) | 66.8 (10.0) | 67.3 (9.6) | 67.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 43 | 142
  Male | 42 | 44 | 49 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 33 | 33 | 107
  Not Hispanic or Latino | 52 | 59 | 59 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 8 | 7 | 22
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 6 | 7 | 3 | 16
  White | 76 | 73 | 78 | 227
  More than one race | 3 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 7 | 3 | 3 | 13
  Brazil | 9 | 7 | 8 | 24
  Colombia | 5 | 4 | 5 | 14
  Germany | 2 | 2 | 0 | 4
  Hungary | 1 | 3 | 0 | 4
  Israel | 7 | 2 | 8 | 17
  Italy | 5 | 2 | 4 | 11
  Mexico | 10 | 11 | 11 | 32
  Poland | 7 | 6 | 8 | 21
  Romania | 2 | 6 | 4 | 12
  Russia | 10 | 8 | 8 | 26
  South Africa | 3 | 2 | 4 | 9
  Spain | 7 | 10 | 11 | 28
  Ukraine | 2 | 8 | 4 | 14
  United States | 16 | 18 | 14 | 48
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.38 (1.06) | 8.28 (1.03) | 8.25 (0.87) | 8.30 (0.99)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 144.72 (15.56) | 143.10 (14.98) | 144.20 (15.10) | 144.01 (15.17)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 26 Comparing Sotagliflozin 400 mg Versus Placebo
Description: An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline to Week 26
Population: Intent-to-treat (ITT) population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data was imputed using the retrieved dropouts & washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 92
percentage of HbA1c | -0.11 (0.151) | -0.40 (0.131)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.0962, ANCOVA; Difference in Least Square (LS) Means = -0.29, 95% CI 2-sided [-0.628 to 0.051], Standard Error of Mean 0.173

2. Secondary Outcome: Change From Baseline in HbA1c at Week 26 Comparing Sotagliflozin 200 mg Versus Placebo
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data was imputed using the retrieved dropouts & washout imputation method.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 200 mg
Number analyzed (Participants) | 93 | 92
percentage of HbA1c | -0.11 (0.151) | -0.07 (0.162)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8124, ANCOVA; Difference in LS Means = 0.05, 95% CI 2-sided [-0.338 to 0.431], Standard Error of Mean 0.196

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 92 | 92
millimole per liter (mmol/L) | 0.069 (0.4482) | -0.291 (0.5056) | -0.644 (0.4348)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline FPG as a covariate; Test type: Superiority; p = 0.5501, ANCOVA; Difference in LS Means = -0.361, 95% CI 2-sided [-1.5431 to 0.8220], Standard Error of Mean 0.6033
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1779, ANCOVA; Difference in LS Means = -0.714, 95% CI 2-sided [-1.7524 to 0.3246], Standard Error of Mean 0.5298

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 92 | 92
kilogram (kg) | 0.39 (0.615) | -0.43 (0.480) | -1.02 (0.490)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline body weight as a covariate; Test type: Superiority; p = 0.2432, ANCOVA; Difference in LS Means = -0.82, 95% CI 2-sided [-2.197 to 0.557], Standard Error of Mean 0.703
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0487, ANCOVA; Difference in LS Means = -1.41, 95% CI 2-sided [-2.810 to -0.008], Standard Error of Mean 0.715

5. Secondary Outcome: Change From Baseline in SBP at Week 12 in Participants With Baseline SBP ≥130 mmHg
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: Analysis population included all participants with baseline SBP ≥130 mmHg in ITT population where, ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data are imputed using control-based copy reference multiple imputation under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 73 | 68 | 73
mmHg | -2.70 (1.815) | -4.84 (1.882) | -7.10 (1.842)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.3954, ANCOVA; Difference in LS Means = -2.14, 95% CI 2-sided [-7.066 to 2.792], Standard Error of Mean 2.515
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0716, ANCOVA; Difference in LS Means = -4.40, 95% CI 2-sided [-9.185 to 0.386], Standard Error of Mean 2.442

6. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data are imputed using control-based copy reference multiple imputation under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 92 | 92
mmHg | -2.50 (1.762) | -5.74 (1.752) | -7.86 (1.794)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 12 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.1232, ANCOVA; Difference in LS Means = -3.24, 95% CI 2-sided [-7.365 to 0.881], Standard Error of Mean 2.103
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0098, ANCOVA; Difference in LS Means = -5.36, 95% CI 2-sided [-9.433 to -1.292], Standard Error of Mean 2.077

7. Secondary Outcome: Percentage Change From Baseline in the Urine Albumin: Creatinine Ratio (UACR) at Week 26 in Participants With Baseline UACR >30 Milligrams Per Gram (mg/g)
Description: An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated.
Time Frame: Baseline to Week 26
Population: Analysis population included all participants with baseline UACR > 30 mg/g in ITT population where, ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures. Missing data was imputed using the retrieved dropouts & washout imputation method.
Measure: Geometric Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 66 | 71 | 75
percent change | -4.56 (NA) — An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated. | -26.99 (NA) — An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated. | -30.66 (NA) — An ANCOVA model was used for analysis. No Measure of Dispersion was pre-specified to be calculated.
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 was analyzed using an ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and log-transformed baseline UACR as a covariate; Test type: Superiority; p = 0.222, ANCOVA; Percent Difference = -20.37, 95% CI 2-sided [-44.75 to 14.77]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.1965, ANCOVA; Percent Difference = -21.17, 95% CI 2-sided [-45.05 to 13.10]

8. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 92 | 92
percentage of participants | 2.2 | 5.4 | 8.7
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Percentage difference between treatment groups using the Cochran-Mantel-Haenszel test stratified by the randomization strata of HbA1c (≤8.5, >8.5%) at screening, randomization strata of metformin use at screening (Yes, No), and the randomization strata of mean SBP (<130, ≥130 mmHg) at screening; Test type: Superiority; p = 0.2420, Cochran-Mantel-Haenszel; Percentage Difference = 3.2, 95% CI 2-sided [-2.17 to 8.66]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0513, Cochran-Mantel-Haenszel; Percentage Difference = 6.5, 95% CI 2-sided [0.04 to 12.93]

9. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26
Time Frame: Week 26
Population: ITT population included all randomized participants, irrespective of compliance with the study protocol and procedures.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 92 | 92
percentage of participants | 4.3 | 16.3 | 17.4
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0066, Cochran-Mantel-Haenszel; Percentage Difference = 12, 95% CI 2-sided [3.48 to 20.61]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel; Percentage Difference = 13, 95% CI 2-sided [4.28 to 21.75]

10. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participants or clinical investigation participants administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the investigational medicinal product (IMP).
Time Frame: First dose of study drug to last dose of study drug (up to 56.3 weeks) + 4 weeks
Population: Safety population included all randomized participants who received at least one dose of double-blind IMP. Two participants were randomized to Sotagliflozin 400 mg and dosed with Sotagliflozin 200 mg and 400 mg treatments during the study. Data for these participants were summarized in the Sotagliflozin 200 mg arm in the safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 94 | 90
percentage of participants | 82.8 | 86.2 | 81.1

11. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤ 70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤ 70 mg/dL].
Time Frame: up to 56.3 weeks
Population: Safety population included all randomized participants who received at least 1 dose of double-blind investigational medicinal product (IMP) (regardless of the amount of treatment administered).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 93 | 94 | 90
percentage of participants
  Any hypoglycemia | 40.9 | 40.4 | 38.9
  Documented symptomatic hypoglycemia | 35.5 | 28.7 | 27.8
  Severe or documented symptomatic hypoglycemia | 35.5 | 30.9 | 27.8

ADVERSE EVENTS:
Time Frame: Deaths: Up to approximately 60 weeks; Adverse Events: First dose of study drug to last dose of study drug (up to 56.3 weeks) + 4 weeks
Description: Safety population included all randomized participants who received at least one dose of double-blind IMP. Hypoglycemia was captured and handled separately from other adverse events and is reported in the outcome measure section.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 6/93 | 6/94 | 3/90
Serious Adverse Events (participants affected / at risk) | 21/93 | 18/94 | 20/90
Other Adverse Events (participants affected / at risk) | 44/93 | 44/94 | 29/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | Sotagliflozin 200 mg (N=94) | Sotagliflozin 400 mg (N=90)
Hypertension (Vascular disorders) | 0 | 1 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Hepatitis C antibody positive (Investigations) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 2 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 2 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=93) | Sotagliflozin 200 mg (N=94) | Sotagliflozin 400 mg (N=90)
Hypertension (Vascular disorders) | 5 | 1 | 3
Glomerular filtration rate decreased (Investigations) | 3 | 10 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 5
Renal impairment (Renal and urinary disorders) | 7 | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 9 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 | 9 | 3
Influenza (Infections and infestations) | 5 | 5 | 2
Nasopharyngitis (Infections and infestations) | 4 | 8 | 1
Urinary tract infection (Infections and infestations) | 16 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03242018/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT03242018/SAP_001.pdf